CLINICAL TRIAL: NCT05301036
Title: Personalized Ultrasonic Brain Stimulation for Depression: A Pilot Study of Target Engagement and Mood Effects
Brief Title: Personalized Ultrasonic Brain Stimulation for Depression
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brian Mickey, Professor of Psychiatry, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00148802
Record Dates: First submitted 2022-03-20; First posted 2022-03-29 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Major Depressive Episode

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation (Experimental): Personalized low-intensity transcranial focused ultrasound stimulation of deep brain target (subgenual cingulate or alternative targets)
  Interventions: Device: Diadem prototype
- Sham stimulation (Sham Comparator): Personalized low-intensity transcranial focused ultrasound stimulation of lateral ventricle
  Interventions: Device: Diadem prototype

INTERVENTIONS:
Device: Diadem prototype — Diadem prototype device delivers personalized low-intensity transcranial focused ultrasound stimulation

SUMMARY:
This study will evaluate a new form of non-invasive brain stimulation for individuals with depression. Personalized low-intensity transcranial focused ultrasound stimulation will first be delivered using a range of stimulation parameters during psychological and physiological monitoring. A well-tolerated stimulation protocol will then be selected for subsequent testing in a blinded randomized sham-controlled cross-over trial to evaluate brain target engagement using magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65, any gender
2. Primary diagnosis of major depressive disorder or bipolar disorder
3. Current moderate-to-severe depressive episode, without psychotic features, lasting at least 2 months
4. Self-rated 16-item Quick Inventory of Depressive Symptomatology (QIDS) total score > 10
5. Stated willingness to comply with all study procedures and avoid changes to psychiatric treatments (medications, psychotherapy) for the duration of the study
6. For females of reproductive potential: negative pregnancy test or use of highly effective contraception for at least 1 month prior to baseline; agreement to use such a method throughout the study
7. Capacity to provide informed consent; provision of a signed and dated consent form

Exclusion Criteria:

1. History of serious brain injury or other neurologic disorder
2. Poorly managed general medical condition
3. Pregnant or breast feeding
4. Implanted device in the head or neck
5. MRI intolerance or contraindication
6. Brain stimulation (e.g., ECT, TMS, VNS) in the past month
7. Suicidal ideation (Columbia Suicide Severity Rating Scale screen item #2, past month)
8. Lifetime history of a serious suicide attempt
9. Moderate-to-severe substance use disorder (past 3 months)
10. Obsessive compulsive disorder (past month)
11. Posttraumatic stress disorder (past month)
12. Schizophrenia-spectrum disorder (lifetime)
13. Neurocognitive disorder (past year)
14. Personality disorder as a current focus of treatment
15. Clinically inappropriate for participation in the study as determined by the study team

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-12-14 (Estimated)

PRIMARY OUTCOMES:
Target engagement: MRI quantification of brain activation | 1 day at MRI study visit
  Blood oxygenation level dependent (BOLD) or arterial spin labeling (ASL) response to active versus sham stimulation
Target engagement: MRI quantification of brain connectivity | 1 day at MRI study visit
  Resting functional connectivity of target in response to active versus sham stimulation
Change in depression severity measured with the HDRS-6 | 1 day and 7 days after stimulation
  6-item Hamilton Depression Rating Scale (HDRS-6), range 0-22, higher score represents greater depression
Change in Sadness scale of PANAS-X | 1 hour, at stimulation study visit
  Positive and Negative Affect Schedule Extended (PANAS-X), range 0-100, higher score represents greater sadness

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Mickey, MD, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riis TS, Feldman DA, Vonesh LC, Brown JR, Solzbacher D, Kubanek J, Mickey BJ. Durable effects of deep brain ultrasonic neuromodulation on major depression: a case report. J Med Case Rep. 2023 Oct 28;17(1):449. doi: 10.1186/s13256-023-04194-4. PMID 37891643